CLINICAL TRIAL: NCT04666987
Title: A Prospective, Non-interventional, Single Arm Study Investigating Long-term Glycaemic Control in Patients With Type 2 Diabetes Initiating Xultophy® (IDegLira) in a Realworld Setting in Italy
Brief Title: A Research Study Looking at Long-term Blood Sugar Control in People With Type 2 Diabetes Being Treated With Xultophy® in a Real-world Setting in Italy
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9068-4740; U1111-1253-1809 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-11-20; First posted 2020-12-14 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec; Liraglutide; IDegLira

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Xultophy®: Participants are patients with Type 2 Diabetes (T2D) treated with Xultophy® (IDegLira) in a real-world setting in Italy
  Interventions: Drug: Insulin degludec and liraglutide (IDegLira)

INTERVENTIONS:
Drug: Insulin degludec and liraglutide (IDegLira) — Paricipants will be treated with commercially available Xultophy® according to routine clinical practice at the discretion of the treating physician, following approved label in Italy. The decision to initiate treatment with commercially available Xultophy® has been made by the patient and the treating physician before and independently from the decision to participate in this study.

SUMMARY:
The purpose of the study is to collect information on how Xultophy® works in patients like them with type 2 diabetes. Participants will get Xultophy® as prescribed to them by the study doctor. The study will last for about 18 months. Participants will be asked questions about their health and diabetes treatment as part of the normal study doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities (study-related activities include any procedure related to recording of data according to the protocol).
* Male or female, age greater than or equal to 18 years at the time of signing informed consent.
* Patient diagnosed with T2D greater than or equal to 12 months prior to signing informed consent.
* The decision to initiate treatment with commercially available Xultophy® has been made by the patient and the treating physician before and independently from the decision to participate in this study.
* Treated with basal insulin with or without use of oral antidiabetics (OADs), with or without use of bolus insulin prior to initiating Xultophy®.
* For patients transferring from a regimen including bolus insulin, upon initiation of Xultophy® the bolus insulin component of the treatment regimen was stopped.
* The patient initiated Xultophy® treatment for at least 2 months, but no more than 3 months prior to signing informed consent.
* Available and documented HbA1c measurement no more than 3 months prior to Xultophy® initiation.

Exclusion Criteria:

* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Diagnosed with type 1 diabetes mellitus, maturity-onset diabetes of the young, latent autoimmune diabetes in adults, gestational diabetes or any hyperglycaemic state other than T2D.
* Women known to be pregnant or breastfeeding, or women planning to become pregnant during the conduct of the study.
* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Participation in another T2D clinical study that involves any clinical intervention or administration of an investigational drug within 3 months prior to enrolment into the study.
* Any contraindications for Xultophy®, including hypersensitivity to the active substances or any of the excipients as specified in the Xultophy® local label.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants are patients with Type 2 Diabetes (T2D) treated with Xultophy® (IDegLira) in a real-world setting in Italy.
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin (HbA1c) | From baseline (V0, month 0) to 6 months after initiation.
  Percent (%) point
  Baseline is defined as the time of Xultophy® initiation (V0); if the endpoint variable is unavailable at (V0), the most recent value within 3 months prior to Xultophy® initiation will be used.
  (This definition of baseline applies to all outcome measures.)

SECONDARY OUTCOMES:
Change in HbA1c | From baseline (V0, month 0) to end of study (V3, 18 ±3 months)
HbA1c levels less than 7% (yes/no) | At end of study (V3, 18 ±3 months)
  Percentage of patients - yes
HbA1c levels less than 7% without hypoglycaemic episodes (yes/no) | At end of study (V3, 18 ±3 months)
  Percentage of patients - yes
Reason for switching to Xultophy® (precoded question list) | At baseline (V0, month 0)
  Percentage of patients
Change in Xultophy® daily dose | From baseline (V0, month 0) to end of study (V3, 18 ±3 months)
  Dose steps/day
Number of self-reported non-severe hypoglycaemia episodes (defined as an episode with symptoms and/or self monitored blood glucose (SMBG) value less than or equal to 3.9 mmol/L) based on recollection | Reported at enrolment (V1 - month 0), intermediate visits (V2.X - 0-17 months) and at end of study (V3, 18 ±3 months). Number of episodes occurring in the 4 weeks prior to study visit
  Number of episodes
Number of self-reported nocturnal nonsevere hypoglycaemic episodes (defined based on the patient's perception of whether or not it was night) based on recollection | Reported at enrolment (V1 - month 0), intermediate visits (V2.X - 0-17 months) and at end of study (V3, 18 ±3 months). Number of episodes occurring in the 4 weeks prior to study visit
  Number of episodes
Number of self-reported severe hypoglycaemic episodes (Defined as an episode of hypoglycaemia requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective action) based on recollection | Reported at enrolment (V1 - month 0), intermediate visits (V2.X - 0-17 months) and at end of study (V3, 18 ±3 months). Number of episodes occurring in the 4 weeks prior to study visit
  Number of episodes
Treatment intensification (addition of prandial insulin, increase in total insulin dose or number of concomitant oral antidiabetics (OADs)) (yes/no) | At end of study (V3, 18 ±3 months)
  Percentage of patients with treatment intensification
Treatment simplification (decrease in insulin dose or number of concomitant OADs) (yes/no) | At end of study (V3, 18 ±3 months)
  Percentage of patients with treatment simplification

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (28):
- Italy (28):
  - Ospedale Santa Maria Goretti - UOD Diabetologia, Latina, LT
  - ICS Maugeri, Pavia, Pv
  - A.O. SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - INRCA, Ancona
  - Azienda Sanitaria Usl Toscana Sud Est - Ospedale San Donato, Arezzo
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - ASST OSpedali Civili ad indirizzo Metabolico Diabetologico, Brescia
  - Centro Polispecialistico Asl Toscana Nord Ovest, Carrara
  - D.S. 43 Casoria Asl Napoli 2 Nord, Casoria
  - H Cannizzaro Malattie endocrine e del ricambio e nutrizione, Catania
  - Ospedale S. Maria del Prato, Feltre
  - A.O.U. Ospedali Riuniti, Foggia
  - Ospedale Camberlingo, Francavilla Fontana
  - Ospedale Policlinico San Martino, Genova
  - A.O.U. Policlinico Martino, Messina
  - ASL Napoli 3 sud, Napoli
  - PSP Loreto Crispi, Napoli
  - Ospedale San Francesco d'Assisi, Oliveto Citra
  - Azienda Ospedaliera Padova, Padua
  - AUSL Pescara, Pescara
  - Ospedale San Jacopo, Pistoia
  - P.O. Praia a Mare ASP Cosenza, Praia a Mare
  - Policlinico Umberto I Clinica Medica DH Diabetologia, Roma
  - Casa della Salute Antistio, Roma
  - Policlinico Universitario AGemelli DH Patologie dell'Obesità, Rome
  - A.O.U. San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Ospedale San Donà di Piave, San Donà di Piave
  - ASUFC Udine, Udine

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com